CLINICAL TRIAL: NCT04049656
Title: A Prospective, Randomized, PACU Blinded, Clinical Utility Study to Confirm the Safety and Efficacy of HFVI-Guided Analgesic Administration in Surgical Subjects Receiving Balanced Sevoflurane-Fentanyl Anesthesia
Brief Title: Confirmatory Study of HFVI Guided Analgesic Administration in Surgical Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Mdoloris Medical Systems (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OCR27162; 20192697 (Other: WIRB)
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-07

CONDITIONS: Analgesia
Keywords: Sevoflurane-Fentanyl Anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: A Prospective, Randomized, PACU Blinded, Clinical Utility Study to Confirm the Safety and Efficacy of HFVI-Guided Analgesic Administration in Surgical Subjects Receiving Balanced Sevoflurane-Fentanyl Anesthesia
Who Masked: Participant, Care Provider
Masking Description: Investigators administering anesthesia will be informed as to whether or not HFVI information will be unmasked to help guide analgesic administration. However, subjects who participate in the trial and the PACU assessors of pain levels will be blinded to study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HFVI intervention group (Experimental): Subjects in the HFVI intervention group will be monitored in the same manner as the control group, but the HFVI monitor display will also be available to the anesthesia provider in real time. Bolus doses of 25ug or 50 ug of fentanyl will be recommended to be administered when the HFVI values begin to decrease below 50, and as needed based on the judgment of the clinician responsible for the case. All anesthetic medications that are given, patient events, and vital sign recordings will be included in the anesthetic record and data collection forms.
  Interventions: Device: HFVI
- Standard of Care Group (No Intervention): Subjects receiving a balanced maintenance anesthetic consisting primarily of a sevoflurane hypnotic (titrated to a BIS range of 40-60) and fentanyl analgesia. Subjects randomized to the control group (Standard Practice) will have analgesia administered as needed according to standard clinical monitoring and practice requirements based on the judgment of the clinician responsible for the case. The HFVI monitor will be applied, but the display will be masked in this control group population.

INTERVENTIONS:
Device: HFVI — Subjects in the HFVI intervention group will be monitored in the same manner as the control group, but the HFVI monitor display will also be available to the anesthesia provider in real time. Bolus doses of 25ug or 50 ug of fentanyl will be recommended to be administered when the HFVI values begin to decrease below 50, and as needed based on the judgment of the clinician responsible for the case. All anesthetic medications that are given, patient events, and vital sign recordings will be included in the anesthetic record and data collection forms.
  Arms: HFVI intervention group

SUMMARY:
The current study is intended to be a prospective clinical performance validation study designed to confirm the clinical utility of HFVI-guided fentanyl administration during sevoflurane anesthesia.

The overall objective of this study is to confirm the safety and efficacy of HFVI-guided analgesic administration in comparison to standard clinical practice. The primary efficacy endpoint will be the amount of postoperative pain reported in the PACU, as measured using a nurse administered Numerical Rating Scale (NRS) pain score.

DETAILED DESCRIPTION:
HFVi was designed to provide a standardized measure of the parasympathetic component (p∑) of the Autonomous Nervous System (ANS). It tracts changes of the p∑ tonus induced by each respiratory cycle (spontaneous or artificial) to measure the relative balance of parasympathetic and sympathetic tone as reflected in the EKG signal.

These rapid changes of the p∑ tonus express themselves at the sinus node level by changes of the time interval separating two R waves of the electrocardiogram. The following normal RR intervals constitute the tachogram (displayed as respiratory pattern on the monitor). The p ∑ component is evaluated after filtering, standardization and re-sampling of the R-R series, by measuring the surface generated by respiratory cycles on the tachogram. Higher p∑ tonus is reflected as a larger measured surface area. In contrast, the measured surface decreases when the p∑ decreases.

HFVi, a measure of the surface area, is expressed in the form of a dimensionless index ranging from 0 to 100. This index reflects the relative activity of the parasympathetic nervous system. It expresses the relative quantity of the present p∑ tonus compared to the Para and sympathetic tonus. The measure of HFVi displayed represents the average of a sequence of measurements: each elementary measure is realized on 64 seconds of data, updated each second using a sliding window.

During development, a probabilistic interpretation of the HFVi was used to relate index values to a clinical state in an anesthetized subject. A significant hemodynamic response (increase of the heart rare or blood pressure of 20% compared to the baseline) within 10 minutes was used as an indicator of nociception/inadequate analgesia.

As a measure of parasympathetic tone, HFVi may be influenced by many factors and thus be difficult to interpret in many of the following situations:

* arrhythmia
* no breathing (ex : apnea due to intubation)
* Respiratory rate lower than 9 cycles/min
* Tidal volume variable on the measuring time, thus 64 seconds
* Irregular breathing (when the patient speaks, laugh or cough)
* pace maker (some types)
* heart transplantation
* Drug use having a significant effect on the sinus cardiac activity

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* American Society of Anesthesiologist Physical Status 1 or 2
* Body Mass Index range of 19-35 kg.m-2.
* Planned spinal or open abdominal surgery expected to last 1-3 hours utilizing a balanced sevoflurane-fentanyl general anesthetic

Exclusion Criteria:

* Subjects are unable or unwilling to give informed consent.
* Emergency surgery
* Women who are currently pregnant or not using a medically acceptable means of birth control
* Cardiac morbidity, including non-regular sinus cardiac rhythm or implanted cardiac pacemaker
* Concurrent medications with a major effect upon the sinus node including prescribed antimuscarinic agents, α2-adrenergic agonists, β1-adrenergic antagonists, and antiarrhythmic agents
* Expected duration of surgery less than 1 hour (60 minutes) or greater than 3 hours (180 minutes)
* Pre-operative chronic opioid use or chronic pain, equivalent to requiring oxycodone 20mg per oral, per day for more than 6 weeks
* Allergy or intolerance to any of the anticipated study medications, such as history of malignant hyperthermia during anesthesia
* Planned use of neuraxial anesthesia
* Clinically significant abnormality or clinically significant unstable medical condition, as indicated by medical history, physical examination, ECG results, or clinical laboratory testing, that in the Investigator's judgment might pose a potential safety risk to the subject or limit interpretation of the trial results, e.g., any uncontrolled thyroid disorders, hepatic, cardiac, pulmonary and renal malfunctioning.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Change in Numerical Pain Scores (NPS) | 15 minutes; 30 minutes; 45 minutes; 60 minutes
  The change in numerical pain scores reported during the first hour (scores at 15, 30, 45, and 60 minutes) of recovery. The NPS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of pain, with 0 being 'no pain' and 10 being 'the worst pain.' Subjects and clinical pain assessors will remain blinded to treatment group assignment.

SECONDARY OUTCOMES:
Percentage of patients minimal pain (NPS < 3) during recovery | Hour 1
  The percent of subjects with minimal pain (NPS < 3) during recovery
Number of opioid analgesics administered in the operating room (OR) and post-anesthesia care unit (PACU). | Hour 1
  The total amounts of opioid analgesics administered in the OR and PACU, respectively.
Incidence of postoperative nausea and vomiting (PONV) in the PACU | Hour 1
  The incidence of significant PONV (emesis) during recovery in the PACU.

CONTACTS AND LOCATIONS:
Overall Officials: Jay W Johansen, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No